CLINICAL TRIAL: NCT01979016
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Investigating the Efficacy, Safety, Serum Concentration and Biomarker Profile of Dupilumab Administered to Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study to Determine the Safety and Effectiveness of Dupilumab for Treatment of Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1307
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Emollients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo qw (Experimental): Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection once weekly (qw) from Week 1 to Week 15.
  Interventions: Drug: Placebo; Other: Background treatment
- Dupilumab 200 mg qw (Experimental): Two subcutaneous injections of Dupilumab 200 milligram (mg) (for a total of 400 mg) as a loading dose on Day 1, followed by a single 200 mg injection qw from Week 1 to Week 15.
  Interventions: Drug: Dupilumab; Other: Background treatment

INTERVENTIONS:
Drug: Dupilumab
  Other Names: REGN668; SAR231893; Dupixent
  Arms: Dupilumab 200 mg qw
Drug: Placebo — Matching placebo
  Arms: Placebo qw
Other: Background treatment — Participants were required to apply stable doses of a topical emollient (moisturizer) twice daily for at least 7 days before the baseline visit and at least 7 days after the baseline visit (day -7 to day 8).
  Other Names: Topical emollient

SUMMARY:
The primary objective of the study was to assess the efficacy of Dupilumab, compared to placebo, in adult patients with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older;
2. Chronic AD that had been present for at least 3 years before the screening visit;
3. Patients with documented recent history (within 6 months before the screening visit) of inadequate response to out-patient treatment with topical medications, or for whom topical treatments were otherwise inadvisable;
4. Willing and able to comply with all clinic visits and study-related procedures.

Exclusion Criteria:

1. Prior participation in a Dupilumab clinical trial;
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives before the baseline visit;
3. The following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, will likely require such treatment(s) during the first 4 weeks of study treatment:

   * Systemic corticosteroids;
   * Immunosuppressive/immunomodulating drugs;
   * Phototherapy for AD;
4. Treatment with topical corticosteroids, tacrolimus and/or pimecrolimus within 1 week before the baseline visit;
5. Treatment with certain biologics;
6. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks before the baseline visit;
7. Planned major surgical procedure during the participant's participation in this study;
8. Participant was a member of the investigational team or his/her immediate family;
9. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit
10. Pregnant or breast-feeding women or women planning to become pregnant or breastfeed during the study;

Note: The information listed above is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial therefore not all inclusion/exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- United States (3):
  - Chicago, Illinois
  - New York, New York
  - Dallas, Texas
- Montreal, Quebec, Canada

REFERENCES:
- [Derived] Callewaert C, Nakatsuji T, Knight R, Kosciolek T, Vrbanac A, Kotol P, Ardeleanu M, Hultsch T, Guttman-Yassky E, Bissonnette R, Silverberg JI, Krueger J, Menter A, Graham NMH, Pirozzi G, Hamilton JD, Gallo RL. IL-4Ralpha Blockade by Dupilumab Decreases Staphylococcus aureus Colonization and Increases Microbial Diversity in Atopic Dermatitis. J Invest Dermatol. 2020 Jan;140(1):191-202.e7. doi: 10.1016/j.jid.2019.05.024. Epub 2019 Jun 25. PMID 31252032
- [Derived] Guttman-Yassky E, Bissonnette R, Ungar B, Suarez-Farinas M, Ardeleanu M, Esaki H, Suprun M, Estrada Y, Xu H, Peng X, Silverberg JI, Menter A, Krueger JG, Zhang R, Chaudhry U, Swanson B, Graham NMH, Pirozzi G, Yancopoulos GD, D Hamilton JD. Dupilumab progressively improves systemic and cutaneous abnormalities in patients with atopic dermatitis. J Allergy Clin Immunol. 2019 Jan;143(1):155-172. doi: 10.1016/j.jaci.2018.08.022. Epub 2018 Sep 5. PMID 30194992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in USA and Canada between 05 December 2013 and 30 January 2015. A total of 66 participants were screened in the study.
Pre-assignment Details: Out of 66 participants, 54 participants were randomized and treated in the study. Participants were randomized in 1:1 ratio to receive Dupilumab 200 mg once weekly (qw) or placebo qw.
Groups:
- Placebo qw: Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 15.
- Dupilumab 200 mg qw: Two subcutaneous injections of Dupilumab 200 mg (for a total of 400 mg) as a loading dose on Day 1, followed by a single 200 mg injection qw from Week 1 to Week 15.
Period: Overall Study
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Started | 27 | 27
Completed | 25 | 26
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo qw | Dupilumab 200 mg qw | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (15.73) | 38.5 (13.55) | 41.3 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 20 | 19 | 39
  Black or African American | 3 | 3 | 6
  Asian | 3 | 5 | 8
  Other | 1 | 0 | 1
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  units on a scale | 34.2 (14.59) | 33.4 (15.41) | 33.8 (14.87)
Investigator Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  units on a scale | 3.5 (0.51) | 3.5 (0.51) | 3.5 (0.50)
Weekly Peak Pruritus Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS was an assessment tool that was used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at worst moment during previous 24 hours (for maximum itch intensity on a scale of 0-10 [0=no itch;10=worst itch imaginable]).
  units on a scale | 7.4 (2.04) | 7.1 (2.42) | 7.3 (2.22)
Global Individual Signs Score (GISS) Total Score [Mean (Standard Deviation); unit: units on a scale] — Individual components of the AD lesions (erythema, infiltration/papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0 = none, 1 = mild, 2 = moderate and 3 = severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
  units on a scale | 8.9 (1.69) | 8.4 (1.82) | 8.6 (1.76)
Patient Oriented Eczema Measure (POEM) Score [Mean (Standard Deviation); unit: units on a scale] — The POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
  units on a scale | 21.4 (5.60) | 21.7 (5.55) | 21.6 (5.52)
Body Surface Area (BSA) Involvement with Atopic Dermatitis [Mean (Standard Deviation); unit: Percentage of BSA] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  Percentage of BSA | 54.5 (26.91) | 53.8 (29.72) | 54.2 (28.08)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: Units on a scale] — SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  Units on a scale | 65.1 (13.36) | 64.2 (17.67) | 64.6 (15.52)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: Units on a scale] — DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL.
  Units on a scale | 14.9 (7.05) | 17.0 (7.67) | 16.0 (7.38)
Total Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: Units on a scale] — The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
  Units on a scale | 12.7 (6.70) | 13.3 (7.66) | 13.0 (7.13)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Eczema Area Severity Index Score (EASI) to Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Values after first rescue medication use were set to missing and missing values imputed by last observation carried forward (LOCF).
Time Frame: Baseline to Week 16
Population: Full analysis set (FAS) population that included all participants who were randomized into this study and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percent change | -5.8 (8.16) | -75.2 (8.15)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a mixed model repeated measures (MMRM) model; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean Difference = -69.4, 95% CI 2-sided [-92.5 to -46.2] — Dupilumab 200 mg qw vs Placebo qw

2. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Values after first rescue medication were set to missing and participants with missing IGA score at Week 16 were considered as non-responders.
Time Frame: Week 16
Population: FAS population was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percentage of participants | 0 | 37.0
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Percentage difference = 37.0, 95% CI 2-sided [18.82 to 55.25] — Dupilumab 200 mg qw vs Placebo qw

3. Secondary Outcome: Percentage of Participants Who Achieved IGA Score Reduction From Baseline of ≥2 Points at Week 16
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Participants with reduction in IGA score from baseline of ≥2 points at Week 16 were reported. Values after first rescue medication were set to missing and participants with missing IGA score at Week 16 were treated as non-responders.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percentage of participants | 3.7 | 51.9
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage difference = 48.1, 95% CI 2-sided [28.00 to 68.30] — Dupilumab 200 mg qw vs Placebo qw

4. Secondary Outcome: Absolute Change From Baseline in Pruritus Numeric Rating Scale (NRS) at Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Values after first rescue treatment were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: Analysis was performed on FAS. Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 26
units on a scale | -0.98 (0.398) | -3.64 (0.405)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.66, 95% CI 2-sided [-3.80 to -1.52] — Dupilumab 200 mg qw vs Placebo qw

5. Secondary Outcome: Percent Change From Baseline in Pruritus Numeric Rating Scale (NRS) at Week 16
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: FAS population. Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 26
percent change | -8.36 (8.098) | -56.44 (8.248)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -48.08, 95% CI 2-sided [-71.31 to -24.85] — Dupilumab 200 mg qw vs Placebo qw

6. Secondary Outcome: Absolute Change From Baseline in EASI Score to Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
units on a scale | -3.7 (2.65) | -25.2 (2.65)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -21.5, 95% CI 2-sided [-29.0 to -14.0] — Dupilumab 200 mg qw vs Placebo qw

7. Secondary Outcome: Absolute Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score to Week 16
Description: SCORAD was a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranged from 0 (absent disease) to 103 (severe disease). Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
units on a scale | -5.1 (3.60) | -36.4 (3.60)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -31.3, 95% CI 2-sided [-41.5 to -21.1] — Dupilumab 200 mg qw vs Placebo qw

8. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score to Week 16
Description: SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS Population was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percent change | -8.2 (5.41) | -54.8 (5.40)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -46.6, 95% CI 2-sided [-62.0 to -31.3] — Dupilumab 200 mg qw vs Placebo qw

9. Secondary Outcome: Percentage of Participants Who Achieved 50%, 75% and 90% Reduction From Baseline in EASI Score ( EASI-50, EASI-75, and EASI-90 Respectively) at Week 16
Description: EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranged from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50, EASI-75 and EASI-90 responders were the participants who achieved ≥50%, ≥75% and ≥90% respectively, overall improvement in EASI score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing EASI score at Week 16 were counted as non-responders.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percentage of participants
  Participants with EASI-50 | 22.2 | 77.8
  Participants with EASI-75 | 14.8 | 66.7
  Participants with EASI-90 | 0 | 33.3
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 50% reduction from baseline in EASI score (EASI-50). Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Percentage difference = 55.6, 95% CI 2-sided [33.38 to 77.73]
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 75% reduction from baseline in EASI score (EASI-75). Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Percentage difference = 51.9, 95% CI 2-sided [29.59 to 74.12]
Statistical Analysis 3: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 90% reduction from baseline in EASI score (EASI-90). Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel; Percentage difference = 33.3, 95% CI 2-sided [15.55 to 51.11]

10. Secondary Outcome: Percentage of Participants Who Achieved 50%, 75% and 90% Reduction From Baseline in SCORAD Score (SCORAD-50, SCORAD-75 and SCORAD-90 Respectively) at Week 16
Description: SCORAD was a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). SCORAD-50, SCORAD-75 and SCORAD-90 responders were the participants who achieved ≥50%, ≥75% and ≥90% respectively, overall improvement in SCORAD score from baseline to Week 16. Values after first rescue treatment were set to missing and participants with missing SCORAD score at Week 16 were counted as non-responders.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percentage of participants
  Participants with SCORAD-50 | 7.4 | 55.6
  Participants with SCORAD-75 | 0 | 11.1
  Participants with SCORAD-90 | 0 | 7.4
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 50% reduction from baseline in SCORAD Score (SCORAD-50). Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Percentage difference = 48.1, 95% CI 2-sided [27.0 to 69.3]
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 75% reduction from baseline in SCORAD Score (SCORAD-75). Analysis was performed by a MMRM model; Test type: Superiority; p = 0.0792, Cochran-Mantel-Haenszel; Percentage difference = 11.1, 95% CI 2-sided [-0.7 to 23.0]
Statistical Analysis 3: Comparison: Placebo qw vs Dupilumab 200 mg qw; Statistical comparison for percentage of participants who achieved 90% reduction from baseline in SCORAD Score (SCORAD-90). Analysis was performed by a MMRM model; Test type: Superiority; p = 0.1573, Cochran-Mantel-Haenszel; Percentage difference = 7.4, 95% CI 2-sided [-2.5 to 17.3]

11. Secondary Outcome: Absolute Change From Baseline in Participant's Oriented Eczema Measure (POEM) Score to Week 16
Description: POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
units on a scale | -2.6 (1.34) | -13.1 (1.37)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -10.4, 95% CI 2-sided [-14.3 to -6.6]

12. Secondary Outcome: Percent Change From Baseline in Participant's Oriented Eczema Measure (POEM) Score to Week 16
Description: POEM was a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
percent change | -12.1 (6.18) | -58.3 (6.31)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Analysis was performed by a MMRM model; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -46.2, 95% CI 2-sided [-63.9 to -28.5]

13. Secondary Outcome: Change From Baseline in Global Individual Signs Score (GISS) Components (Erythema, Infiltration/Papulation, Excoriations, and Lichenification) to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0 = none, 1 = mild, 2 = moderate and 3 = severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).Values after first rescue medication use were set to missing and missing values were imputed by LOCF.
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
units on a scale
  Change in Erythema GISS | 0.0 (0.14) | -0.7 (0.14)
  Change in Infiltration/Papulation GISS | -0.1 (0.13) | -1.0 (0.13)
  Change in Excoriation GISS | -0.3 (0.14) | -1.3 (0.14)
  Change in Lichenification GISS | -0.1 (0.14) | -1.2 (0.14)

14. Secondary Outcome: Changes From Baseline in GISS Cumulative Score to Week 16
Description: as for outcome 13
Time Frame: Baseline to Week 16
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 200 mg qw
Number analyzed (Participants) | 27 | 27
units on a scale | -0.5 (0.46) | -4.2 (0.46)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 200 mg qw; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -3.7, 95% CI 2-sided [-5.02 to -2.39]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 32) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events: AEs that developed/worsened during the on treatment period (time period from the administration of first dose of study drug to the final visit [Week 32]).
Groups:
- Placebo qw: Participants exposed to Placebo (for Dupilumab) (mean exposure of 10 weeks).
- Dupilumab 200 mg qw: Participants exposed to Dupilumab 200 mg qw (mean exposure of 14 weeks).
Arm/Group | Placebo qw | Dupilumab 200 mg qw
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27 | 0/27
Other Adverse Events (participants affected / at risk) | 17/27 | 20/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qw (N=27) | Dupilumab 200 mg qw (N=27)
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo qw (N=27) | Dupilumab 200 mg qw (N=27)
Conjunctivitis allergic (Eye disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Injection site erythema (General disorders) | 1 | 2
Injection site reaction (General disorders) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 5 | 3
Post procedural infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 4
Viral upper respiratory tract infection (Infections and infestations) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 | 4
Dermatitis Infected (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.